CLINICAL TRIAL: NCT00461695
Title: Influence of Persistent CMV-infection on Immune Senescence Evaluated With a Prospective Vaccination Trial Against Tick-borne Encephalitis Virus in Healthy Elderly Individuals (CYTEL-Study)
Brief Title: Influence of Persistent CMV-infection on Immune Senescence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Division of Infectious Diseases and Hospital Epidemiology (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CYTEL-Protocol V1.A1
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Immune Senescence
Keywords: Cytomegalovirus (CMV); Tick-borne encephalitis virus (TBEV); Ageing; Vaccine; Immunity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CMV-seropositive (Other): Cytomegalovirus-seropositive individuals at screening (week 0). Intervention: Intervention: Vaccination against tick-borne encephalitis by intramuscular injection into the left (or right) deltoid muscle of 0.5 ml FSME Immun CC for adults (2.4 ug of formalin inactivated TBEV antigen) at time point 0, after 4 weeks and after 24 weeks.
  Interventions: Biological: Vaccination against TBEV (FSME Immun CC)
- CMV-seronegative (Other): Cytomegalovirus-seronegative individuals at screening (week 0). Intervention: Vaccination against tick-borne encephalitis by intramuscular injection into the left (or right) deltoid muscle of 0.5 ml FSME Immun CC for adults (2.4 ug of formalin inactivated TBEV antigen) at time point 0, after 4 weeks and after 24 weeks.
  Interventions: Biological: Vaccination against TBEV (FSME Immun CC)

INTERVENTIONS:
Biological: Vaccination against TBEV (FSME Immun CC) — Intramuscular injection into the left (or right) deltoid muscle of 0.5 ml FSME Immun CC for adults (2.4 ug of formalin inactivated TBEV antigen) at time point 0, after 4 weeks and after 24 weeks.

SUMMARY:
Recent studies indicate that persistent viral infections particularly with Cytomegalovirus (CMV) might have a negative impact on immune senescence (i.e. immunocompetence of elderly individuals). We will test this hypothesis by performing a vaccination trial in healthy elderly individuals subdivided in two groups of CMV-seropositive and CMV-seronegative individuals. All individuals will be vaccinated with the currently licensed vaccine for the prevention of TBE (FSME Immun CC) which is recommended for the general population in our area. Vaccination efficacy will be monitored longitudinally concerning the TBEV-specific antibody (TBEV-neutralization, TBEV-specific ELISA) and T cell response (ELISpot, cytokine production).

Vaccination efficacy will be compared between CMV+ and CMV- individuals and correlated with the CMV-specific immune response in CMV+ individuals.

ELIGIBILITY:
Inclusion criteria:

* Age > 70 years
* Healthy according to a health questionnaire (completed before screening)
* TBE-Vaccination indicated (exposure to TBEV-infested ticks possible)
* Capable to make an informed decision and to understand the informed consent form
* Informed consent signed by patient and study physician

Exclusion criteria:

* Previous exposure to TBEV (natural or vaccination)
* Immunodeficiency, history of autoimmune disease or current intake of immune-modulating drugs (corticosteroids a.s.o.)
* Persistent (> 3 months) pharmacological treatment with more than one drug of relevance (exception: combination antihypertensives)
* Contraindication for TBEV-vaccination
* Condition that would drastically interfere with clinic attendance and/or adherence to the protocol
* Past medical history or current treatment for one of the following conditions: Chronic cardiac disease (Coronary heart disease, heart failure), chronic pulmonary disease (COPD), chronic kidney disease, diabetes mellitus, previous stroke, epilepsy, Parkinsons disease, dementia
* Hemoglobin <12 g/l
* Random plasma glucose (RPG) > 11.1 mmol/l OR fasting plasma glucose (FPG) > 6.9 mmol/l (FPG required, if RPG is 7.0-11.0 mmol/l)
* Calculated Creatinin-Clearance < 50 ml/min
* TBEV-serology positive

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 183 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of anti-TBEV-antibodies measured by TBEV-neutralisation assay and ELISA one month after each TBEV-vaccine administration in the group of CMV-seropositive versus CMV-seronegative individuals | One month after each TBEV-vaccine administration

SECONDARY OUTCOMES:
Efficacy of TBEV-vaccination in healthy elderly individuals (Geometric mean antibody titer measured by TBEV-neutralisation test). | One month after 3rd TBEV-vaccine administration
Safety of TBEV-vaccination in healthy elderly individuals. | One month after 3rd TBEV-vaccine administration.

CONTACTS AND LOCATIONS:
Overall Officials: Urs Karrer, MD, Principal Investigator — University Hospital Zurich, Department of Infectious Diseases and Hospital Epidemiology
Locations (1):
- University Hospital Zurich, Department of Infectious Diseases and Hospital Epidemiology, Zurich, Switzerland